CLINICAL TRIAL: NCT06359795
Title: Exploring the Value of 18F-AlF-FAPI PET/CT in Assessing the Activity of Thyroid Eye Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FAPI-TED
Record Dates: First submitted 2024-04-07; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Thyroid Eye Disease
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Patients with TED will be recruited in the study.
  Interventions:
  Diagnostic Test: 18F-AlF-FAPI PET/CT and 99mTc-DTPA SPECT/CT.
  Interventions: Diagnostic Test: 18F-AlF-FAPI PET/CT, 99mTc-DTPA SPECT/CT

INTERVENTIONS:
Diagnostic Test: 18F-AlF-FAPI PET/CT, 99mTc-DTPA SPECT/CT — Patients underwent 18F-AlF-FAPI PET/CT and 99mTc-DTPA SPECT/CT scans within 10 days.

SUMMARY:
FAPI PET has been developed as a promising approach for the evaluation of fibroinflammatory, such as in inflammatory bowel disease. This prospective study aims to explore the value of 18F-AlF-FAPI PET/CT in assessing the activity of Thyroid Eye Disease (TED) and investigate whether FAPI PET/CT may be superior to 99mTc-DTPA SPECT/CT for the diagnosis, therapy response assessment, and follow-up of TED.

DETAILED DESCRIPTION:
Subjects with TED underwent 18F-AlF-FAPI PET/CT and 99mTc-DTPA SPECT/CT for activity assessment within a 10-day period. On 18F-AlF-FAPI PET/CT, uptake in the extraocular muscles was quantified using SUV metrics and target-to-background ratio. On 99mTc-DTPA SPECT/CT, uptake in the extraocular muscles was semi-quantified using the uptake ratio. Activity of TED was determined through comprehensive clinical data. The correlation between SUV metrics and activity status was calculated to explore the value of 18F-AlF-FAPI PET/CT in assessing TED activity. The diagnostic accuracy of 18F-AlF-FAPI PET/CT and 99mTc-DTPA SPECT/CT in assessing TED activity was compared. Additionally, the correlation of changes in SUV metrics and therapy response will be calculated to explore the value of 18F-AlF-FAPI PET/CT in therapy response assessment of TED.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Patients diagnosed with TED;
3. Complete understanding and voluntary participation in this study, with the signing of an informed consent form.

Exclusion Criteria:

1. Severe liver or kidney dysfunction;
2. Inability to maintain a supine position for 5 minutes to cooperate with the examination;
3. Suffering from claustrophobia or other psychiatric disorders;
4. Patients planning pregnancy or in the prenatal or lactation period;
5. Other conditions deemed unsuitable for participation in the trial by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | through study completion, an average of 6 months
  The accuracy of 18F-AlF-FAPI PET/CT in assessing the activity of TED.

SECONDARY OUTCOMES:
The value to predict therapy response | through study completion, an average of 12 months
  The changes of SUV metrics on 18F-AlF-FAPI PET/CT to predict therapy response
Diagnostic accuracy comparison | through study completion, an average of 6 months
  Comparing the diagnostic accuracy in assessing the activity of TED activity between 18F-AlF-FAPI PET/CT and 99mTc-DTPA SPECT/CT.
FAPI expression and SUV metrics | through study completion, an average of 12 months
  Correlation between SUV metrics on PET and FAPI expression in patients with surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Li, Dr., Principal Investigator — Peking University Third Hospital
Locations (1):
- Dept. of Nuclear Medicine, Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No